CLINICAL TRIAL: NCT02482064
Title: A Clinical Comparative Study of Two Types of Maxillary Obturators Made of Heat Cure Acrylic Resin or Flexible Resin
Brief Title: Using Flexible Resin in Maxillary Obturators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-RemPro-01-2015
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Patients Who Had Undergone Partial or Complete Maxillectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional Obturators (No Intervention): Patients will use traditional obturators which are going to be made from ordinary heat-activated acrylic resin.
- Flexible Obturators (Experimental): Patients will use the new obturators made from flexible resin.
  Interventions: Other: Flexible resin

INTERVENTIONS:
Other: Flexible resin — This material 'Flexible resin' is going to be used in the construction of the 'flexible obturators'.
  Arms: Flexible Obturators

SUMMARY:
Ten patients who had had maxillectomy will be assigned to two groups employing two types of 'temporary obturators. The obturators in the first group will be made from heat cure acrylic resin, whereas those in the second group from flexible resin.

A comparison will be made between the two materials in terms of oral-nasal seal using the drinking water test as well as the mirror test.

DETAILED DESCRIPTION:
Oral rehabilitation following partial maxillectomy presents numerous clinical and technical issues. Using soft-tissue undercuts in the palatal side of the upper jaw is so useful for prostheses' retention over and above the abutment teeth. The use of flexible materials can serve this aim. The current study aims to compare the efficacy of nasal-oral seal using flexible materials against the traditional method of using heat activated acrylic materials.

ELIGIBILITY:
Inclusion Criteria:

* patient who had partial or complete maxillectomy
* two weeks should have passed at least before being included in the study.
* patient should have completed their radiotherapy.

Exclusion Criteria:

* patients under the age of 10 years
* patients who had had their operations more than five months before the being recruited.
* patients who are under radiotherapy when asked to participate in the study.

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Amount of leaking water drops from the nose | 30 minutes following appliance insertion in the mouth
  Each patient is asked to drink an amount of water and keep a specific amount of water in the mouth for two to three minutes. He/she is asked to rotate his/her head 20-30 degrees downward and forward. During this period the amount of leaking water drops from the nose is collected and weighted.
Amount of air flow through the nose during speech | 30 minutes following appliance insertion in the mouth
  Each patient is asked to utter the following letters: K, T, D. A cold small mirror is placed in front of the nose during the utterance of these consonants. If a fogginess is observed on the mirror, this means that there is an oral-nasal leakage of air.

CONTACTS AND LOCATIONS:
Overall Officials: Huda Yahia, DDS, Principal Investigator — MSc student, Removable Prosthodontic Department, University of Damascus Dental School; Eyad Al-Shaarani, DDS MSc PhD, Study Director — Professor of Removable Prosthodontics, University of Damascus Dental School
Locations (1):
- Department of Removable Prosthodontics, University of Damascus Dental School, Damascus, Rif-dimashq Governorate, Syria

REFERENCES:
- [Background] Aramany MA. Basic principles of obturator design for partially edentulous patients. Part II: Design principles. 1978 [classical article]. J Prosthet Dent. 2001 Dec;86(6):562-8. doi: 10.1067/mpr.2001.121619. No abstract available. PMID 11753303
- [Background] Grossmann Y, Savion I. The use of a light-polymerized resin-based obturator for the treatment of the maxillofacial patient. J Prosthet Dent. 2005 Sep;94(3):289-92. doi: 10.1016/j.prosdent.2005.06.014. PMID 16126082
- [Background] MacCarthy D, Murphy N. Replacement of an obturator section of an existing two-piece implant-retained edentulous obturator. J Prosthet Dent. 2000 Jun;83(6):652-5. PMID 10842133
- [Background] Kanazawa T, Yoshida H, Furuya Y, Shimodaira K. Sectional prosthesis with hollow obturator portion made of thin silicone layer over resin frame. J Oral Rehabil. 2000 Sep;27(9):760-4. doi: 10.1046/j.1365-2842.2000.00584.x. PMID 11012850